CLINICAL TRIAL: NCT00242476
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, 16-Week Study to Assess the Effect of Vitamin D3 8400IU Once Weekly on Body Sway and Neuromuscular Function in Men and Women Aged 70 Years or Older
Brief Title: A Study to Assess the Effectiveness of an Investigational Drug in Elderly Subjects With Low Vitamin D Levels (0822A-009)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0822A-009; MK0822A-009; 2005_089
Record Dates: First submitted 2005-10-18; First posted 2005-10-20 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0822A

SUMMARY:
This study will assess the effectiveness of an investigational drug in elderly subjects with low vitamin D levels.

ELIGIBILITY:
Inclusion Criteria:

* Man or a woman 70 years old or older in general good health

Exclusion Criteria:

* Having any form of neurological impairments that may impair motor function.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 216 (Actual)
Dates: Start 2005-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Mediolateral body sway at 16 weeks. | at 16 weeks

SECONDARY OUTCOMES:
Functional status assessed using the Short Physical Performance Battery Test determined at 16 weeks. General safety and tolerability at 16 weeks. | at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Lips P, Binkley N, Pfeifer M, Recker R, Samanta S, Cohn DA, Chandler J, Rosenberg E, Papanicolaou DA. Once-weekly dose of 8400 IU vitamin D(3) compared with placebo: effects on neuromuscular function and tolerability in older adults with vitamin D insufficiency. Am J Clin Nutr. 2010 Apr;91(4):985-91. doi: 10.3945/ajcn.2009.28113. Epub 2010 Feb 3. PMID 20130093